CLINICAL TRIAL: NCT01220141
Title: Prospective Observational Study on NovoSeven® Room Temperature Stable (VII25) in Patients With Haemophilia A or B
Brief Title: Observational Study on Safety of Room Temperature Stable NovoSeven® in Patients With Haemophilia A or B
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN7025-3601; U1111-1116-2012 (Other: WHO)
Record Dates: First submitted 2010-10-12; First posted 2010-10-13 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-04

CONDITIONS: Congenital Bleeding Disorder; Haemophilia A; Haemophilia B
MeSH Terms: conditions — Hemophilia A; Hemophilia B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A
  Interventions: Drug: activated recombinant human factor VII

INTERVENTIONS:
Drug: activated recombinant human factor VII — Administration of room temperature stable NovoSeven® (activated recombinant human factor VII) in dosages prescribed by the treating physician according to the product labelling text approved in his country.

SUMMARY:
This study is conducted in Europe and Asia. The aim of this observational study is to monitor antibody formation towards the room temperature stable formulation of NovoSeven® (activated recombinant human factor VII).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with congenital haemophilia A or B with inhibitors to factor VIII or factor IX
* Treated with room temperature stable NovoSeven®

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male patients with haemophilia A or B with inhibitors treated with room temperature stable NovoSeven® (activated recombinant human factor VII).
Sampling Method: Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2010-11; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Reduced therapeutic response and neutralising antibodies to activated recombinant human factor VII as confirmed by central laboratory | after 25 exposure days

SECONDARY OUTCOMES:
Adverse events reported as potentially related to activated recombinant human factor VII | after 25 exposure days

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (14):
- Prov. de Buenos Aires, Argentina
- Vienna, Austria
- Brussels, Belgium
- Paris La Défense Cedex, France
- Mainz, Germany
- Budapest, Hungary
- Tehran, Iran
- Dublin, Ireland
- Rome, Italy
- Warsaw, Poland
- Paço de Arcos, Portugal
- Bratislava, Slovakia
- Malmo, Sweden
- Crawley, United Kingdom

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com